CLINICAL TRIAL: NCT06224387
Title: A Multi-center, Open-label, Dose Escalation/Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of CTS2190 in Patients With Solid Tumors
Brief Title: CTS2190 Phase I /II Clinical Study in Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CytosinLab Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTS2190-CI01
Record Dates: First submitted 2023-05-07; First posted 2024-01-25 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumors; Pancreatic Cancer; Non-small Cell Lung Cancer; Triple-negative Breast Cancer
Keywords: Phase I/II; pharmacodynamic; Pharmacokinetics; Tolerability
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: QD and durg holiday,PO.
Masking Description: QD and durg holiday,PO.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation/Dose Expansion (Experimental): 4-6 dose groups are pre-specified in Dose Escalation,and 4 arms in Dose Expansion.
  Interventions: Drug: CTS2190 capsules

INTERVENTIONS:
Drug: CTS2190 capsules — 4-6 dose groups are pre-specified in Dose Escalation,and 4 arms in Dose Expansion.
  Other Names: CTS2190

SUMMARY:
This is a first in human study in patients with advanced or metastatic solid tumors. The first part of the study is an open-label, dose escalation and the second part is an open label dose expansion in specific tumor types. The study drug, CTS2190, is a PRMT1 inhibitor administered orally. The study is planned to treat up to 224 participants.

DETAILED DESCRIPTION:
This is a Phase 1/2 multi-center, open label study in solid tumor patients. Phase 1（Part1) is a dose escalation study of oral CTS2190 in patients with solid tumors，which is planned to treat up to 144 participants.

Phase 2（Part2) is an open label, dose expansion study in specific tumor types. In both parts of the study, participants who tolerate the drug may continue the treatment until disease progression.

The study duration for each subject is defined as beginning from 28 days prior to the first dose, until the subject withdrawal of informed consent, end of treatment, loss to follow-up or death, completes 48 weeks of continuous treatment or the study ends early, whichever occurs first. The end of study is defined as the date when the last subject completes the last visit specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria can be included in this study:

1. Male or female ≥ 18 years of age at signing of ICF.
2. Part 1: histologically or cytologically confirmed locally advanced or metastatic solid tumors at screening who cannot be treated surgically and have failed standard treatment (PD during treatment or after the last treatment) recommended by the current clinical diagnosis and treatment standards or guidelines, or cannot tolerate standard treatment, or refuse standard treatment and/or currently have no effective treatment available.

   Part 2: histologically or cytologically confirmed advanced solid tumors (including pancreatic cancer, non-small cell lung cancer and/or other tumors, such as gastric cancer, colorectal cancer, etc.) at screening who cannot be treated surgically and have failed standard treatment (PD during treatment or after the last treatment) recommended by the current clinical diagnosis and treatment standards or guidelines, or cannot tolerate standard treatment, or refuse standard treatment and/or currently have no effective standard treatment available.
3. At least one measurable tumor lesion at screening [according to RECIST V1.1 criteria (see appendix 1)].
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 (Appendix 2) at screening.
5. With a life expectancy ≥ 12 weeks at screening.
6. With good organ function at screening, including:

   * Liver function: total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN) (if the following conditions occur, isolated bilirubin >1.5 × ULN is acceptable if: bilirubin is fractionated and direct bilirubin <35%, or the patients is diagnosed with Gilbert syndrome), alanine aminotransferase (ALT) ≤ 2.5 × ULN, and aspartate aminotransferase (AST) ≤ 2.5 × ULN (for patients with liver metastases or tumor infiltration, the criteria can be relaxed to TBIL ≤ 1.5 × ULN, ALT ≤5 × ULN, and AST ≤ 5 × ULN);
   * Renal function: blood creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min [calculate the creatinine clearance using Cockcroft-Gault formula (appendix 3)];
   * Hematology: platelet ≥ the lower limit of the laboratory normal range, and absolute neutrophil count (ANC) ≥ 1.5 × 109/L, and hemoglobin ≥ 100 g/dL;
   * Cardiac function: QT interval corrected by Fridericia method (QTcF) ≤ 450 ms (male) or ≤ 470 ms (female) (see the appendix 3 for calculation formula).
   * Coagulation function: International normalized ratio (INR) ≤ 1.5 × ULN, or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
7. Female patients of non-childbearing age or female patients of childbearing age who have negative pregnancy test results and promise to take sufficient and effective contraceptive measures or adhere to abstinence from the screening period to 90 days after the last administration, or male patients who promise to take sufficient and effective contraceptive measures or adhere to abstinence from the screening period to 90 days after the last administration (see the appendix 4). Patients are not allowed to donate sperm within 6 months from the start of administration to 6 months after the end of investigational drug administration.
8. Patients who understand and voluntarily signs the ICF, are willing to and able to complete the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

Subjects should not participate in this clinical study if any of the following conditions is met:

1. Female patients in pregnancy or lactation.
2. Patients with dysphagia.
3. Patients who cannot tolerate venipuncture or have a history of syncope judged by the investigator to be clinically significant.
4. Uncontrolled tumor-related pain.
5. Allergic or intolerant to the active ingredients or excipients of the investigational drug judged by the investigator.
6. Treatment with radiotherapy for the target lesion within 4 weeks before the first administration of the investigational drug, or accepted any anti-tumor drugs/ treatments (including but not limited to chemotherapy, targeted therapy, immunotherapy) within 5 half-lives before the first administration of the investigational drug, whichever is longer; or patients who have received herbal therapies with anti-tumor indications within 1 week before the first administration.
7. Primary central nervous system (CNS) tumor or CNS metastasis at screening. The following patients can be considered for enrollment: after treatment and being stable for ≥ 3 months, patients who have completed the treatment at least 10 days before the start of the study treatment; the corticosteroid treatment has been terminated for ≥ 5 days when the study treatment starts, the neurological function is stable, and it is estimated that no steroids or antiepileptic drugs will be required during the study treatment.
8. Patients judged by the investigator to have uncontrolled pleural effusion, pericardial effusion, or peritoneal effusion (requiring repeated drainage, multiple times a month or more frequently) at screening. Allow patients to indwell catheters regardless of drainage frequency.
9. Patients with untreated or clinically symptomatic spinal cord compression that has not been controlled (except for patients who have received treatment and have stable symptoms, whose imaging examination shows that they are stable for at least 4 weeks before the first administration, and who have no evidence of brain edema and do not require glucocorticoid treatment).
10. Patients with ≥ 2 malignant tumors within 5 years before the first administration. Except for cured early-stage malignancies (carcinoma in situ or stage I tumor), such as adequately treated cervical carcinoma in situ, basal cell or squamous epithelial cell skin cancer.
11. Patients who are found to have active pulmonary tuberculosis infection within 1 year before enrollment through medical history, or those with a history of active pulmonary tuberculosis infection more than one year ago who have not received formal treatment.
12. Interstitial lung disease or interstitial pneumonia, including clinically significant radiation pneumonia (i.e., affecting activities of daily living or requiring intervention).
13. Severe infection within 4 weeks before the first administration, including but not limited to bacteremia and severe pneumonia, etc. requiring hospitalization; CTCAE ≥ grade 2 active infection requiring systemic antibiotic treatment within 2 weeks before the first administration.
14. History of serious cardiovascular and cerebrovascular diseases, including but not limited to serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, degree II-III atrioventricular block, etc.; acute coronary syndrome, congestive cardiac failure, aortic dissection, stroke or other grade 3 or above cardiovascular and cerebrovascular events within 6 months before the first administration; New York Heart Association (NYHA) cardiac function classification (see appendix 5) ≥ grade II or left ventricular ejection fraction (LVEF)<50% or hypertension that cannot be clinically controlled (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg).
15. Positive hepatitis B virus surface antigen (HBsAg) and the number of copies of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) ≥ 500 IU/mL (or 2500 copies, or the lower limit of the positive detection value of the study site) at screening, HBsAg (-), hepatitis B core antibody (HBcAb) (+) and the number of copies of HBV DNA≥ 500 IU/mL (or 2500 copies, or the lower limit of the positive detection value of the study site) after treatment of HBV infection, or positive hepatitis C antibody (HCVAb) and hepatitis C virus (HCV) ribonucleic acid (RNA) ≥ ULN of the study site; those with a history of liver cirrhosis (Child Pugh class B or C) or active syphilis infection.
16. Patients who have active diseases or a history of autoimmune diseases that may relapse (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.) at screening, except patients suffering clinically stable autoimmune thyroid disorder.
17. History of immunodeficiency, including HIV positive, or those suffering from other acquired or congenital immunodeficiency diseases, or with a history of allograft. Autotransplantation should be completed at least 3 months before screening.
18. Those who had clinically significant hemorrhage symptoms within 3 months before the first administration. Patients who significantly coughed up blood within 4 weeks before the first administration of the investigational drug, and the amount of hemoptysis each time reached half a teaspoon (2.5 mL) or more; patients who had arterial/venous thrombosis events within 6 months before the first administration, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism, central retinal vein occlusion (RVO), etc.; those who are receiving anticoagulant treatment at the time of screening; patients with potential thrombosis or at the risk of coagulation judged by the investigator.
19. Patients who have received other unlisted clinical investigational drugs or treatments within 4 weeks (or 5 drug half-lives, whichever is longer) before the first administration.
20. Patients who have used live vaccine or attenuated vaccine within 4 weeks before the first administration, or plan to use live vaccine or attenuated vaccine during the study period.
21. Patients who have used potent cytochrome enzyme (CYP)3A4 inhibitors or inducers within 2 weeks before the first administration, or need to use potent CYP3A4 inhibitors or inducers until 7 days after the last dose (see the appendix 6).
22. Major surgery (except for surgery for diagnostic purposes) within 4 weeks before the first administration, or expected to undergo major surgery (except for surgery for diagnostic purposes) during the study period, or have undergone diagnostic or minimally invasive surgery within 7 days before the first administration.
23. Adverse reactions from previous anti-tumor treatment have not recovered to ≤ CTCAE V5.0 grade 1 (except for alopecia and grade 2 neurotoxicity caused by chemotherapy drugs, grade 2 hypothyroidism caused by anti-tumor treatments, hypertension and other toxicities that are judged to have no safety risks by the investigator).
24. Patients who are judged by the investigator to have a history of other serious systemic diseases, or not suitable for participating in the trial for any other reason (the patient has mental illness, alcohol abuse, drug use or drug abuse that may affect his/her compliance with the trial or may interfere with the interpretation of the study results).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation：The maximum tolerated dose (MTD) | During the DLT observation period: 25 days after the first administration
  The MTD is defined as the dose level at which the DLT rate is closest to the target toxicity incidence (i.e., 0.3) during the DLT observation period (within 25 days after the first administration).
Dose Escalation：The recommended phase 2 dose (RP2D) | During the DLT observation period: 25 days after the first administration
  The recommended phase 2 dose (RP2D) of CTS2190 Based on the review of all available data including, but not limited to, safety, tolerability, PK, PD and preliminary anti-tumor activity, RP2D may be determined.
Dose Expansion：Objective response rate(ORR) | Every 6 weeks for the duration of study participation.
  The percentage of participants having complete response (CR) or partial response (PR))assessed based on RECIST V1.1.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) characteristics:Peak concentration(Cmax) | Day1 to Day 4 Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  Peak concentration of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics: time to peak concentration (Tmax) | Single-dose stage: Day1 to Day 4; Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day1.
  time to peak concentration of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：area under concentration-time curve from zero to infinity (AUC0-∞) | Single-dose stage: Day 1 to Day 4, Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 D 16, Cycle 3 Day 1 and Cycle 5 Day 1
  area under concentration-time curve from zero to infinity of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：area under concentration-time curve from zero to time of the last detectable concentration (AUC0-t) | single-dose stage: Day 1 to Day 4
  area under concentration-time curve from zero to time of the last detectable concentration of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：elimination half-life (T1/2) | single-dose stage: Day 1 to Day 4
  elimination half-life (T1/2) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：apparent clearance (CL/F) | single-dose stage: Day 1 to Day 4
  apparent clearance (CL/F) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：apparent volume of distribution (Vz/F) | single-dose stage: Day 1 to Day 4
  apparent volume of distribution (Vz/F) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：mean residence time (MRT) | single-dose stage: Day 1 to Day 4
  mean residence time (MRT) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：area under concentration-time curve from time of the last administration to the last detectable concentration (AUC0-t,ss) | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  area under concentration-time curve from time of the last administration to the last detectable concentration (AUC0-t,ss) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：area under concentration-time curve from time of last administration to infinity (AUC0-∞,ss) | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  area under concentration-time curve from time of last administration to infinity (AUC0-∞,ss) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：time to steady-state peak concentration (Tmax, ss) | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  time to steady-state peak concentration (Tmax, ss) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：steady-state peak concentration (Cmax,ss) | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  steady-state peak concentration (Cmax,ss) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：steady-state trough concentration (Css trough) | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  steady-state trough concentration (Css trough) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：steady-state elimination half-life (T1/2, ss) | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  steady-state elimination half-life (T1/2, ss) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：steady-state elimination rate constant (λz,ss) | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  steady-state elimination rate constant (λz,ss) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：steady-state apparent clearance (CL/F,ss) | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  steady-state apparent clearance (CL/F,ss) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：steady-state apparent volume of distribution (V/F,ss) | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  steady-state apparent volume of distribution (V/F,ss) of CTS2190 in patients with solid tumors
Pharmacokinetic (PK) characteristics：accumulation indexes Rac,Cmax and Rac,AUC | Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 3 Day 1 and Cycle 5 Day 1
  accumulation indexes Rac,Cmax and Rac,AUC of CTS2190 in patients with solid tumors
Dose Expansion：Objective response rate (ORR) | Every 6 weeks for the duration of study participation
  Objective response rate (ORR) assessed based on the Response Evaluation Criteria in Solid Tumors (RECIST) V1.1.
Incidence of TEAEs and SAEs | Baseline through 28 days after end of treatment, estimated up to 48 weeks
  Before and after treatment, clinically significant changes in vital signs, physical examination, laboratory tests, 12-lead ECG and other safety measures.
Duration of response (DOR) | Every 6 weeks for the duration of study participation
  Duration of response (DOR) assessed based on the Response Evaluation Criteria in Solid Tumors (RECIST) V1.1.
Disease control rate (DCR) | Every 6 weeks for the duration of study participation
  disease control rate (DCR) assessed based on the Response Evaluation Criteria in Solid Tumors (RECIST) V1.1.
Progression-free survival (PFS) | Every 6 weeks for the duration of study participation
  progression-free survival (PFS) assessed based on the Response Evaluation Criteria in Solid Tumors (RECIST) V1.1.
Pharmacodynamic (PD) characteristics of CTS2190 : asymmetric dimethylarginine (ADMA) | Single-dose stage:Day 1; Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day1, Cycle 1 Day 8, Cycle 1 Day 15 and Cycle 3 Day 1
  To explore the changes of asymmetric dimethylarginine (ADMA) in blood of patients with solid tumors before and after administration of CTS2190 and their correlation with the efficacy of CTS2190.
Pharmacodynamic (PD) characteristics of CTS2190 : monomethyl arginine (MMA) | Single-dose stage:Day 1; Multiple-dose stage: Cycle 1 (each cycle is 21 days) Day 1, Cycle 1 Day 8, Cycle 1 Day 15 and Cycle 3 Day 1
  To explore the changes of monomethyl arginine (MMA) in blood of patients with solid tumors before and after administration of CTS2190 and their correlation with the efficacy of CTS2190.

CONTACTS AND LOCATIONS:
Overall Officials: Wu H P, Docotor, Study Chair — CytosinLab Therapeutics Co., Ltd.
Locations (2):
- China (2):
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No